CLINICAL TRIAL: NCT02839460
Title: A Single-Center, Prospective Study to Evaluate Biomarkers of Skeletal Muscle Atrophy in Sarcopenia
Brief Title: A Prospective Study Of Biomarkers Of Skeletal Muscle Atrophy
Acronym: TWEAK
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: TWEAK
Record Dates: First submitted 2016-07-18; First posted 2016-07-21 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Muscle biopsy samples may be retained for mRNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- subjects with sarcopenia: Screening Procedures (Physical Exam, Height & Weight, Vitals, Medical History, CHAMPS, DXA Scan, Physical Performance Testing, Muscle Strength Testing, Blood Collection)
  Day 1 (target +/- 2 days) Outpatient Muscle Biopsy (Vitals, Blood Collection, Muscle Biopsy, update Concomitant Therapy and Procedure-Related AEs/SAEs)
  Day 14 (target +/- 2 days) Safety Follow-up Visit (Vitals, Blood Collection, update Concomitant Therapy and Procedure-Related AEs/SAEs)
  Interventions: Procedure: Outpatient Muscle Biopsy
- healthy, physically-active controls: Screening Procedures (Physical Exam, Height & Weight, Vitals, Medical History, CHAMPS, DXA Scan, Physical Performance Testing, Muscle Strength Testing, Blood Collection)
  Day 1 (target +/- 2 days) Outpatient Muscle Biopsy (Vitals, Blood Collection, Muscle Biopsy, update Concomitant Therapy and Procedure-Related AEs/SAEs)
  Day 14 (target +/- 2 days) Safety Follow-up Visit (Vitals, Blood Collection, update Concomitant Therapy and Procedure-Related AEs/SAEs)
  Interventions: Procedure: Outpatient Muscle Biopsy

INTERVENTIONS:
Procedure: Outpatient Muscle Biopsy — Outpatient Muscle Biopsy involving skeletal muscle sample collected from the vastus lateralis muscle

SUMMARY:
This is a single center, prospective biomarker study to evaluate serum levels of TWEAK and expression levels of TWEAK and Fn14 in muscle biopsies from patients with sarcopenia as well as healthy, physically active controls.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, all candidates must meet the following eligibility criteria at Baseline or at the time point specified in the individual eligibility criterion listed:

All Participants

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information in accordance with national and local subject privacy regulations

Subjects with Sarcopenia

1. Men and postmenopausal women of 65 years of age or older
2. Gait speed measured over 4 meters of <1.0 m/s OR grip strength < 26 kg for men or < 16 kg for women.
3. Appendicular skeletal muscle adjusted for BMI by DXA ≤ 0.789 for men and ≤ 0.512 for women.
4. Weigh at least 40kg;
5. Self-reported difficulty climbing 10 steps OR walking outside on level ground for 1/4 mile

Healthy Controls

1. Men and postmenopausal women of 65 Years of age or older
2. Body mass index (BMI) between 18.5 and 30 kg/m2 inclusive at the time of Screening
3. Measures of Physical Performance and Lean Mass exceed thresholds defined for Sarcopenia group.
4. ≥ 150 minutes/week moderate-intensity physical activity OR regular engagement in resistance training ≥ 2 days/week
5. Willing to maintain a consistent diet and pattern of physical activity for the duration of the study

Exclusion Criteria:

Candidates will be excluded from study entry if any of the following exclusion criteria exist at Screening:

1. History of human immunodeficiency virus (HIV), hepatitis B or C, or tuberculosis (TB)
2. Immunocompromized subjects, as determined by the Investigator, based on medical history, physical examination, or laboratory testing, or due to prior or current immunosuppressive or immunomodulating treatment, including, but not limited to, HIV infection, history of organ transplantation, and anti-rejection therapy
3. Acute infection (urinary, respiratory, other) within past week or hospitalization within one month
4. Participation in any interventional clinical study within 12 weeks
5. A lower limb fracture in the past 6 months or any impairment or disease severely affecting gait (e.g. stroke with hemiparesis, myasthenia gravis, Parkinson's disease, peripheral polyneuropathy, intermittent claudication in advanced peripheral vascular disease, spinal stenosis, or severe osteoarthritis of the knee or hip);
6. Any underlying muscle disease including active myopathy or muscular dystrophy.
7. Confirmed diagnosis of heart failure classified as New York Heart Association Class III and IV (e.g. cardiomyopathy) or hypertrophic cardiomyopathy.
8. Type I diabetes or uncontrolled Type 2 diabetes (HA1C ≥ 9).
9. Requires regular assistance from another person for general activities of daily living (e.g. bathing, dressing)
10. Moderate to Vigorous Exercise performed in week prior to study visits (temporary exclusion - will be rescheduled)
11. Any other condition judged by the Principal Investigator or Study Physician to preclude safe participation in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Subjects over age 65 Subjects with Sarcopenia Subjects who are healthy, physically-active controls
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-11; Primary Completion 2018-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Serum concentration of TWEAK at day 1 | Day 1

SECONDARY OUTCOMES:
Relative expression levels of TWEAK mRNA in muscle biopsy at day 1 | Day 1
Relative expression levels of Fn14 mRNA in muscle biopsy at day 1 | Day 1
Correlation between serum TWEAK levels and muscle strength | Day 1
Incidence of AEs and SAEs | Screening through Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Anton, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Institute on Aging, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No